CLINICAL TRIAL: NCT00059735
Title: A Phase II Study of E7070 in Patients With Progressive Inoperable and/or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: A Safety, Tolerability and Efficacy Study of E7070 in Patients With Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7070-A001-206
Record Dates: First submitted 2003-05-05; First posted 2003-05-07 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Kidney Neoplasms; Carcinoma, Renal Cell; Adenocarcinoma, Renal Cell
Keywords: kidney cancer; kidney neoplasms; renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: E7070

SUMMARY:
The purpose of this study is to determine if E7070 is a safe and effective treatment for cancer of the kidneys.

DETAILED DESCRIPTION:
Renal Cell Carcinoma (RCC) accounts for approximately 2% of all cancers and its incidence is increasing with worldwide deaths of over 100,000 patients per year. About 50% of RCC patients have inoperable or metastatic disease that surgery cannot be performed on. RCC is also considered to be resistant to both radiotherapy and cytotoxic chemotherapy. The purpose of this study is to evaluate the safety and effectiveness of E7070 by assessing progression free survival, tumor response rate, duration of response/stable disease, and survival time. E7070 will be administered as a single iv infusion over 60 minutes on Day 1 of each cycle. Patients will continue treatment with E7070 until they no longer have clinical benefit and have disease progression, or toxicity leads to patient withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old.
* Have histologically/cytologically confirmed clear cell RCC.
* Previously untreated or one prior treatment with immunotherapy (one prior treatment may be represented by single agent interferon, single agent interleukin-2 or a combination of interferon with interleukin-2 with or without accompanying hematological growth factors).
* Documented evidence of progressive disease in the previous 3 months. In the absence of radiographic studies, patients may be entered on the study if they have clinical evidence of progressive disease.
* Have at least one unidimensional measurable lesion of RCC according to the RECIST guidelines. The following will not qualify as measurable lesions: bone, leptomeningeal disease, ascites, pleural/pericardial effusion, lymphangitis cutis/pulmonis, abdominal masses that are not confirmed and followed by imaging techniques, and cystic lesions.
* Be ambulatory and have a Karnofsky performance status >=70%.
* Have a life expectancy of at least 3 months.
* Give written informed consent prior to any study-specific screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
* Be willing and able to comply with the study protocol for the duration of the study.

Exclusion Criteria:

* Woman who are pregnant or breastfeeding. Women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate contraceptive measures (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Fertile male subjects not willing to use contraception and whose female partners are not under adequate contraceptive protection.
* Known CNS metastases (if clinical suspicion of CNS metastases exists appropriate imaging must be performed prior to study entry).
* Prior treatment with chemotherapy (there is no restriction on prior epidermal growth factor directed therapy).
* Severe and uncontrolled cardiac or cardiovascular abnormalities.
* Severe uncontrolled intercurrent infections.
* Subjects with organ allografts.
* Any of the following abnormal screening hematological values: Hemoglobin (Hb) <9g /dL (6 mmol/L), Neutrophils <1.5 x 10^9/L, Platelets <100 x 10^9/L.
* Blood transfusions or growth factors to aid hematological recovery within 2 weeks prior to starting study treatment.
* Any of the following abnormal screening liver function tests: serum bilirubin >= 1.5 x upper normal limit (ULN), alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) >= 2.5 x ULN (unless related to liver metastases in which case >= 5 x ULN).
* The following abnormal screening renal function tests: either a serum creatinine > 1.5 x ULN or a creatinine clearance (estimated from serum creatinine) < 40 mL/minute.
* Prior radiotherapy (except palliative).
* Participation in any investigational drug study or immunotherapy within 4 weeks preceding treatment start.
* History of hypersensitivity to sulphonamides.
* Any concurrent or previous malignancy of a different tumor type within 5 years of starting E7070 treatment except for adequately treated non-melanoma skin cancer or cervical intra-epithelial neoplasia.
* Significant disease, which in the Investigator's opinion would exclude the patient from the study.
* Surgically resectable metastatic disease.
* Legal incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-05; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Yule, MRCP, PhD, Study Director — Eisai Limited
Locations (4):
- United States (3):
  - Sacramento, California
  - New York, New York
  - The Bronx, New York
- Villejuif, France

REFERENCES:
- See also: Related Info — http://www.eisai.com